CLINICAL TRIAL: NCT00333333
Title: Mechanism of Thrombocytopenia in Small for Gestational Age Infants Versus Infants With Maternal Preeclampsia Exposure
Brief Title: Mechanism of Thrombocytopenia in Infants
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: The Cardeza Foundation for Hematologic Research (Other)
Responsible Party: Kelly Zook, MD, Christiana Hospital
Other Study IDs: CCC# 26075
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Thrombocytopenia; Small for Gestational Age (SGA); Preeclampsia
Keywords: Thrombocytopenia; Small for Gestational Age (SGA); Preeclampsia
MeSH Terms: conditions — Thrombocytopenia; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cord blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SGA infants: Infants who are thought to be small for gestational age (SGA)
  Interventions: Procedure: Cord blood
- Pre-eclampsia exposed: Infants who are born to mothers who had pre-eclampsia
  Interventions: Procedure: Cord blood

INTERVENTIONS:
Procedure: Cord blood — Cord blood will be obtained at the time of delivery.

SUMMARY:
This research project is studying the causes for low platelet levels in preterm infants. Platelets are a component of blood that helps with clotting. The purpose of this study is to determine whether the cause for low platelet levels is the same in infants who are born to mothers with preeclampsia and infants who are small for gestational age.

DETAILED DESCRIPTION:
Thrombocytopenia is a common entity in infants who are born to mothers with preeclampsia and in infants who are small for gestational age. There have been several theories to the mechanism underlying thrombocytopenia in these groups of patients. One mechanism suggests that thrombocytopenia in these populations may be secondary to underproduction of platelets. Other studies have implied that low platelet levels may be due to endothelial activation causing platelet consumption. This study is being performed to help determine the mechanism causing thrombocytopenia in infants born to mothers with preeclampsia and comparing it to the mechanism of thrombocytopenia in infants who are small for gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are less than 34 weeks gestation
* Infants born to mothers with preeclampsia
* Infants who are born small for gestational age whose mother did not have preeclampsia

Exclusion Criteria:

* Infants who are greater than 34 weeks gestation
* Infants with known congenital anomalies or known congenital infections

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In utero infants who are small for gestational age or who are exposed to maternal pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine the mechanism of thrombocytopenia in small for gestational age infants versus infants with maternal preeclampsia exposure | Each infant will only be enrolled during the time of birth until cord blood is collected.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Zook, MD, Principal Investigator — Christiana Care Health Systems; Thomas Jefferson University Hospital
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States